CLINICAL TRIAL: NCT05837845
Title: A Randomized Trial to Compare MDMA-assisted Cognitive Processing Therapy (aCPT) Versus a VA Standard-of-care CPT for the Treatment of Severe Posttraumatic Stress Disorder Among Veterans
Brief Title: MDMA-assisted Cognitive Processing Therapy Versus Cognitive Processing Therapy for Veterans With Severe Posttraumatic Stress Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Patricia Suppes (Other)
Collaborators: Stanford University (Other); VA Palo Alto Health Care System (U.S. Federal Agency); Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor-Investigator, Patricia Suppes, Professor, Palo Alto Veterans Institute for Research
Organization: Palo Alto Veterans Institute for Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUP0023APR
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: PTSD
Keywords: MDMA-assisted Therapy; Cognitive Processing Therapy; Veterans; Posttraumatic stress disorder; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: This is a randomized study. Participants will be 1:1 randomized to receive either MDMA-aCPT or CPT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDMA-assisted Cognitive Processing Therapy (MDMA-aCPT) (Experimental): This arm consists of 8-15 virtual CPT sessions (average of 12), one 90-minute, non-drug Preparatory Session, three Experimental Sessions with MDMA (~8 hours), and three 90-minute, non-drug Integration Sessions, occurring over a 9-15-week Treatment Period. Standardized homework is assigned at each CPT session to promote the practice of the skills taught in the session. Participants will receive 80mg MDMA HCl for the first Experimental Session and will have the option of a supplemental dose of 40mg MDMA HCI 1.5-2 hours after the initial dose. For the second and third Experimental Sessions, participants will receive either 80mg or 120mg MDMA HCl as the initial dose, and an optional supplemental dose of 40mg or 60mg MDMA HCl 1.5-2 hours after the initial dose. Participants interested in receiving CPT treatment alone after study completion will have the option to be referred to their local VA PTSD Clinical Team for services 6 months after all study visits are completed.
  Interventions: Drug: MDMA; Behavioral: MDMA-assisted Cognitive Processing Therapy (MDMA-aCPT)
- Cognitive processing therapy (Experimental): This arm consists of 8-15 virtual CPT treatment sessions lasting approximately 1-1.5 hours, occurring over a ~12-16-week Treatment Period. These sessions will take place approximately one week apart. Standardized homework is assigned at each session to promote the practice of the skills taught in the session. Participants will have the option to crossover to the MDMA-aCPT arm 6 months after all study visits are completed.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Drug: MDMA — Participants will receive a flexible divided-dose of MDMA HCl plus therapy at three Experimental Sessions, as well as non-drug Preparatory and Integration Sessions
  Arms: MDMA-assisted Cognitive Processing Therapy (MDMA-aCPT)
Behavioral: Cognitive Processing Therapy — Participants will receive 8-15 (average of 12) sessions of Cognitive Processing Therapy
  Arms: Cognitive processing therapy
Behavioral: MDMA-assisted Cognitive Processing Therapy (MDMA-aCPT) — Participants assigned to MDMA-aCPT will undergo a therapeutic approach administered by trained therapists. MDMA seems to engender internal awareness that even painful feelings that arise are an important part of the therapeutic process. MDMA can elicit feelings of empathy, love, and deep appreciation, along with a clearer perspective of the trauma as a past event, a more accurate perspective about its significance, and a heightened awareness of the support and safety that exists in the present. A combined treatment of MDMA and therapy may be especially useful for treating PTSD because MDMA can attenuate the fear response of a perceived threat to one's emotional integrity and decrease defensiveness without blocking access to memories or preventing a deep and genuine experience of emotion.
  Arms: MDMA-assisted Cognitive Processing Therapy (MDMA-aCPT)

SUMMARY:
In partnership with the Veterans Affairs (VA) Palo Alto Health Care System and Stanford University, this study aims to evaluate clinical outcomes, assess implementation feasibility, and health economics of MDMA-assisted Cognitive Processing Therapy (MDMA-aCPT) in the treatment of posttraumatic stress disorder (PTSD). Through a randomized comparison of MDMA-aCPT versus Cognitive Processing Therapy (CPT), a VA gold standard treatment for PTSD, the proposed study will set the stage for understanding the potential use and application of MDMA-aCPT for PTSD within the VA system.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a serious debilitating disorder that negatively impacts a person's daily life, and can result in diminished cognitive and psychosocial functioning, fractured relationships, inability to maintain employment, substance use disorders, high-cost healthcare utilization, increased depression, and suicide risk. People who suffer from PTSD relive their traumatic experience(s) through nightmares and flashbacks, have difficulty sleeping, and feel detached or estranged. Symptoms can be severe and long lasting.

Many available PTSD treatments, including medications and therapy, effectively treat only a fraction of people who try them. This indicates a need to assess treatments targeting durable remission of PTSD. An extensive list of medications, namely antipsychotics, anxiolytics, antidepressants, and sleep aids, are frequently prescribed off-label but are minimally effective in reducing PTSD symptoms.

Cognitive Processing Therapy (CPT) is a cognitively-oriented approach to treating PTSD developed in the late 1980's by Dr. Patricia Resick. Significant research on CPT has been conducted in the VA system nationally. Across a number of studies, a meta-analysis found the number of subjects that no longer meet PTSD criteria after receiving a full course of CPT ranged from 30% to 97%, and 51% of subjects receiving CPT achieved loss of diagnosis compared to waitlist, self-help booklets, and treatment as usual control groups. There are various task forces and active efforts to deploy CPT more broadly in the VA.

MDMA-assisted cognitive processing therapy (MDMA-aCPT) is a novel treatment package that combines standard CPT with the administration of MDMA (3,4-methylenedioxymethamphetamine) during medication sessions separate from CPT sessions. This includes the regular course of 8-15 CPT sessions, three sessions during which MDMA is used, and an additional one 'preparatory' session and three 'integration' sessions without the use of medication. Data from a series of Phase 2 and Phase 3 studies of MDMA-assisted therapy provide preliminary evidence suggesting that chronic PTSD symptoms are improved by up to three sessions of MDMA-assisted therapy and associated non-drug preparatory and integrative therapy sessions.

Our goal is to learn how MDMA-aCPT compares to CPT in reducing PTSD symptoms among Veterans. Comparing MDMA-aCPT and CPT for the treatment of PTSD is particularly important due to the urgent need for effective treatments within the VA system.

PTSD carries a high public burden, both economically and socially, by increased healthcare utilization, use of social services, lost wages, and disability payments. Given the chronicity of PTSD, low treatment compliance evidenced by high dropouts, and limited recovery with current medications contributing to serious outcomes, PTSD patients exhibit an unmet medical need. Currently, the VA serves approximately nine million Veterans and the conservative estimate of those with PTSD is 25%, or over two million Veterans. The potential importance and benefits of this novel treatment to Veterans, doctors, researchers, and the VA system cannot be underestimated. The clinical effectiveness, implementation evaluation, and economic assessment conducted in this study will provide critical information and understanding of the feasibility of utilization in the VA system.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Are at least 18 years at the time of signing the informed consent
2. Are a U.S Military Veteran
3. Are receiving services from VA Palo Alto Healthcare System, VA San Francisco Healthcare System, or VA NorCal Healthcare System
4. Are fluent in speaking and reading in English
5. Agree to have study visits audio and/or video recorded
6. If assigned to MDMA-aCPT, able to identify appropriate support person(s) to stay with the participant on the evenings of the MDMA sessions
7. Meet DSM-5 criteria for PTSD with a symptom duration of at least 6 months
8. Have severe PTSD symptoms in the last month
9. Body weight of at least 48 kilograms (kg)
10. Is not pregnant, planning to get pregnant, or breastfeeding
11. Capable of giving signed informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful
2. Have current unstable medical illness
3. Have cardiac conditions, including uncontrolled hypertension, prolonged QTc interval, and other cardiac conditions
4. Have received Electroconvulsive Therapy (ECT), ketamine-assisted therapy, or used ketamine within 12 weeks of enrollment
5. Moderate or severe alcohol or cannabis use disorder within the last 12 months
6. Active illicit drug (other than cannabis) or prescription drug substance use disorder at any severity within the last 12 months
7. Have current serious suicide risk
8. Unable or unwilling to stop or safely taper off prohibited medications
9. Have used MDMA (ecstasy) ever
10. Currently enrolled in any clinical study
11. Personal history of primary psychotic disorder, type I bipolar disorder, severe personality disorder, eating disorder with compensatory behaviors, or depressive disorder with psychotic features
12. Lack social support, or lack a stable living situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale (CAPS-5) Total Severity Score | From Baseline to approximately 4 months post-baseline
  The Primary Outcome measure will be the change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score from Baseline to 4 months post-baseline assessed by a blinded study staff rater.
  The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.

SECONDARY OUTCOMES:
Change in Quality of Life Enjoyment and Satisfaction Questionnaire | From Baseline to approximately 4 months post-baseline
  The secondary outcome measure will be the change in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF).
  The Q-LES-Q-SF is a self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. The summary scores were found to be reliable and valid measures of these dimensions in a group of depressed outpatients. The Q-LES-Q-SF measures were related to, but not redundant with, measures of overall severity of illness or severity of depression within this sample. These findings suggest that the Q-LES-Q-SF measures may be sensitive to important differences among depressed patients that are not detected by the measures usually employed. Each item uses a 5-point scale ranging from 1 (very poor) to 5 (very good). The total score ranges from 0-70, with higher scores indicating greater life satisfaction and enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Suppes, MD, PhD, Principal Investigator — VA Palo Alto Healthcare System / Stanford University; Shannon Wiltsey Stirman, PhD, Principal Investigator — VA Palo Alto Healthcare System / Stanford University
Locations (1):
- VA Palo Alto Health Care System / Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No